CLINICAL TRIAL: NCT04939623
Title: Novel Use of Probenecid to Alleviate Symptoms of Opioid Withdrawal in People with Chronic Pain Undergoing Voluntary Opioid Tapering: a Pilot Study
Brief Title: Novel Use of Probenecid to Alleviate Symptoms of Opioid Withdrawal
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Probenacid 1.0
Record Dates: First submitted 2020-09-11; First posted 2021-06-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain; Drug Dependence of Morphine Type; Symptom, Withdrawal
MeSH Terms: conditions — Chronic Pain; Substance Withdrawal Syndrome | interventions — Probenecid

STUDY DESIGN:
Intervention Model Description: 40 participants will be randomized in a 2:2:1 ratio to one of:
  1. Probenecid 500 mg PO BID (16 participants)
  2. Probenecid 1000 mg PO BID (16 participants)
  3. Placebo PO BID (8 participants)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be sequentially randomized. Allocation will be concealed through use of a computer-generated algorithm employing simple randomization without stratification. Participants and the research team will be blinded to group assignment. Randomization will utilize a 2:2:1 ratio (500 mg Probenecid:1000mg Probenecid: placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Probenecid 500 mg PO BID (Active Comparator): Probenecid 500 mg X 1 PO BID and Placebo X 1 PO BID
  Interventions: Drug: Probenecid
- Probenecid 1000 mg PO BID (Active Comparator): Probenecid 500mg X 2 PO BID
  Interventions: Drug: Probenecid
- Placebo PO BID (Placebo Comparator): Placebo X 2 PO BID
  Interventions: Drug: Probenecid

INTERVENTIONS:
Drug: Probenecid — The Investigators aim to recruit 40 participants who will be followed for 12 weeks in duration. Participants will be randomized in a 2:2:1 ratio to one of probenecid 500 mg, 1000 mg, or placebo PO BID for 12 weeks. Justification for use of a non-active placebo comparator includes the fact that this trial is meant to identify tolerability and safety of probenecid in a population of patients living with chronic pain, this will be best measured by comparing to a non-active placebo.
  Other Names: 4-(Dipropylsulfamoyl)benzoic acid; Benemid; Probalan

SUMMARY:
The proposed clinical trial will address the problem of opioid withdrawal. Opioids are essential for pain-relief in the short term, but their continued use is associated with a host of adverse effects. People living with chronic pain who were initiated on opioid therapy now find themselves with a major life-changing problem - dependence on opioid medications. Opioid withdrawal symptoms are a key barrier to decreasing or stopping their opioid medication. Currently, there are few medications that ameliorate the symptoms of opioid withdrawal. This problem is a major part of the opioid crisis in Canada, and impacts people across all demographics and socioeconomic status. A misconception is that only individuals with opioid use disorder are susceptible to opioid withdrawal; on the contrary, appropriate use of prescription opioids to manage pain can lead to significant symptoms of opioid withdrawal when it is reduced or stopped. Patients in Alberta who are at risk for opioid withdrawal, either from prescribed use or misuse will be primarily impacted by this trial.

The investigators have recently explored the underlying causes of opioid withdrawal and identified an important target in the spinal cord that is responsible for producing withdrawal symptoms in rats and mice. The target, a protein called pannexin-1 (Panx1), is located throughout the body, specifically in the brain and spinal cord. Using sophisticated biochemical, genetic, and pharmacological techniques, the investigators demonstrated how Panx1 on immune cells is implicated in the production of opioid withdrawal symptoms after cessation of fentanyl and morphine in opioid dependent rodents. The investigators then attenuated these symptoms of withdrawal using probenecid, a drug which inherently blocks Panx1 activity. Because probenecid is a safe and clinically available drug, the findings could be immediately translated into clinical therapy to support people who are struggling with the symptoms of opioid withdrawal and provide clinicians with a safe and effective option for caring for this population.

DETAILED DESCRIPTION:
The proposed clinical trial will address the problem of opioid withdrawal. Opioids are essential for pain-relief in the short term, but their continued use is associated with a host of adverse effects. People living with chronic pain who were initiated on opioid therapy now find themselves with a major life-changing problem - dependence on opioid medications. Opioid withdrawal symptoms are a key barrier to decreasing or stopping their opioid medication. Currently, there are few medications that ameliorate the symptoms of opioid withdrawal. This problem is a major part of the opioid crisis in Canada, and impacts people across all demographics and socioeconomic status. A misconception is that only individuals with opioid use disorder are susceptible to opioid withdrawal; on the contrary, appropriate use of prescription opioids to manage pain can lead to significant symptoms of opioid withdrawal when it is reduced or stopped. Patients in Alberta who are at risk for opioid withdrawal, either from prescribed use or misuse will be primarily impacted by this trial.

Our team has recently explored the underlying causes of opioid withdrawal and identified an important target in the spinal cord that is responsible for producing withdrawal symptoms in rats and mice. The target, a protein called pannexin-1 (Panx1), is located throughout the body, specifically in the brain and spinal cord. Using sophisticated biochemical, genetic, and pharmacological techniques, the investigators demonstrated how Panx1 on immune cells is implicated in the production of opioid withdrawal symptoms after cessation of fentanyl and morphine in opioid dependent rodents. The investigators then attenuated these symptoms of withdrawal using probenecid, a drug which inherently blocks Panx1 activity. Because probenecid is a safe and clinically available drug, the findings could be immediately translated into clinical therapy to support people who are struggling with the symptoms of opioid withdrawal and provide clinicians with a safe and effective option for caring for this population.

Probenecid was initially developed in the early 1950s as a tool to enhance the activity of penicillin and allow for outpatient treatment of various infections. It increases plasma levels and the half-life of weak organic acids (penicillins, cephalosporins, or other beta-lactam antibiotics) by competitively inhibiting their renal tubular secretion. As a result, it became widely used in combination with beta-lactam antibacterial agents. It is still occasionally used today in combination with cefazolin for the treatment of skin and soft tissue infections, and in combination with cefoxitin or doxycycline as an option for outpatient treatment of pelvic inflammatory disease.

Probenacid also competitively inhibits active reabsorption of uric acid at the level of the proximal convoluted tubule promoting excretion of uric acid, thereby reducing serum urate concentrations.

Probenecid is also used in combination with cidofovir for the prevention of cidofovir-related nephrotoxicity when used to treat cytomegalovirus retinitis in patients with HIV. More recently, the effects of probenecid on serotonin levels and TRPV2 channels has led to speculation about its utility in depression, Parkinson's Disease, and congestive heart failure.

The drug is no longer commercially available in Canada but is commercially available as 500 mg tablets in the United States which can be acquired through Health Canada's Special Access Program. Probenecid can, however, be prepared in Canada by compounding pharmacies.

The study is a single centre, randomized, double blind, placebo-controlled, 12-week clinical trial meant to study probenecid use among adult participants living with chronic non-cancer pain using opioid drug therapy on a daily basis and planning to voluntarily reduce their dose.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with chronic pain. Age greater than or equal to 18 years on the day of enrolment.
2. Subjects are currently taking a daily opioid pain medication and planning to taper the dose.
3. Participants complete at least one voluntary opioid dose reduction in the twelve-week study period.
4. Glomerular filtration rate (GFR) > 50 mL/min
5. Capable of providing informed consent

Exclusion Criteria:

1. Allergy to probenecid or related drugs
2. History of uric acid renal calculi, if known to be urate calculi. If unknown type, then any history of renal calculi.
3. Known G6PD deficiency
4. Active gout in any joint
5. Current use of drugs whose exposure may be prolonged, or risk of toxicity increased when used in combination with probenecid:

   1. Penicillins, specifically ampicillin, penicillin G sodium, and piperacillin
   2. Carbapenems, specifically doripenem and meropenem
   3. Lorazepam, midazolam, nitrazepam
   4. Ketorolac
   5. Oseltamivir
   6. Methotrexate
   7. Mycophenolate
6. Current use of drugs which may mask symptoms of withdrawal:

   a. Clonidine, lofexidine, tizanidine
7. Current use of drugs which may diminish the effect of probenecid:

   a. High dose salicylates including greater than 325 mg PO daily of acetylsalicylic acid (ASA)
8. Pregnancy or breastfeeding
9. Any major comorbid medical condition which might impair follow-up or result in a safety risk to the participant
10. Participation in another clinical trial investigating a drug, medical device, or a medical procedure during the 30 days prior to enrolment.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate tolerability of oral probenecid in patients undergoing voluntary opioid tapering | 12 weeks
  Tolerability will be assessed through use of the "SAFTEE-SI questionnaire recorded as a percentage for each of the three group assignments and again in two groups titled "probenecid" and "placebo".
  Statistical comparisons will be made between groups with regard to the percentage of participants experiencing any given adverse event. (example: rash occurred at a rate of 0% with placebo, 2% with probenecid 500 mg, and 4% with probenecid 1000 mg). Comparisons will also be made between the "probenecid group" and "placebo group" (Example: Blurred vision occurred at a rate of 2% with placebo compared to 4% with probenecid)
To evaluate acceptability of oral probenecid in patients undergoing voluntary opioid tapering | 12 weeks
  Acceptability will be measured by assessing the Percent of patients achieving 80% compliance in each group as measured by returned supply in medication vials.
To evaluate safety of oral probenecid in patients undergoing voluntary | 12 weeks
  Safety will be assessed by the clinical research team who have diagnosed the adverse events which will be recorded as a percentage for each of the three group assignments and again in two groups titled "probenecid" and "placebo".
  Statistical comparisons will be made between groups with regard to the percentage of participants experiencing any given adverse event. (example: rash occurred at a rate of 0% with placebo, 2% with probenecid 500 mg, and 4% with probenecid 1000 mg). Comparisons will also be made between the "probenecid group" and "placebo group" (Example: Blurred vision occurred at a rate of 2% with placebo compared to 4% with probenecid)

SECONDARY OUTCOMES:
To evaluate the feasibility of treatment with probenecid in a patient-directed opioid tapering protocol, in the setting of an interdisciplinary pain clinic | 3 years
  To evaluate the feasibility of treatment with probenecid in a patient-directed opioid tapering protocol, in the setting of an interdisciplinary pain clinic. The sample size of enrolling 40 subjects over a 3 year period will be be used to evaluate the feasibility of a larger study using a similar protocol.
To evaluate whether Panx1 gene variants correlate with opioid withdrawal severity and response to probenecid by collecting salivary samples and performing DNA extraction in a small cohort. | 3 years
  A summary of association analyses between subjects DNA samples will be evaluated to determine PANX1 genetic variants and then analyzed for corellation with the study endpoints (e.g. adverse events, opioid withdrawal) and then be reported by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Montgomery, MD, Principal Investigator — University of Calgary
Locations (1):
- Richmond Road Diagnostic and Treatment Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1 Beyer, R. H., Wiebelhaus, V. D., Russe, H. F., Peck, H. M., & McKinney, S. E. (1950). Benemid: An anticatabolite; its phar- macological properties. Federation Proceedings, 9, 258.
- [Background] Probenecid CPhA Monograph. RxTx. Date of Revision: November 2017. Accessed online at https://www.e-therapeutics.ca on February 21, 2018.
- [Background] Robbins N, Koch SE, Tranter M, Rubinstein J. The history and future of probenecid. Cardiovasc Toxicol. 2012 Mar;12(1):1-9. doi: 10.1007/s12012-011-9145-8. PMID 21938493
- [Background] Benuryl Tablets, Probenecid Tablets. Prescribing Information. Montreal, Quebec. Valeant Canada LP. Date of Revision: September 1, 2004.